CLINICAL TRIAL: NCT05049044
Title: Observational Prospective Study of Quality of Life in Unresectable TNM Stage III NSCLC (OBSTINATE)
Acronym: OBSTINATE
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: GFPC 06-2019
Record Dates: First submitted 2020-11-13; First posted 2021-09-17 (Actual); Last update posted 2025-08-04 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small-cell lung cancer; Unresectable; Advanced stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (10):
- Cohort 1: cRT-CT+IO: Concomitant radio-chemotherapy and consolidation immunotherapy (cRT-CT+IO)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 2: sRT-CT+IO: Sequential radio-chemotherapy and consolidation immunotherapy (sRT-CT+IO)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 3: cRT-CT: Concomitant radio-chemotherapy (cRT-CT)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 4: sRT-CT: Sequential radio-chemotherapy (sRT-CT)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 5: CT: Chemotherapy only (CT)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 6: CT+IO: Chemotherapy plus immunotherapy (CT+IO)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 7: RT: Radiation therapy only (RT)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 8: IO: Immunotherapy only (IO)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 9: TT: Targeted therapy only (TT)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)
- Cohort 10: BSC: Best supportive care only (BSC)
  Interventions: Other: Quality of Life Questionnaire-Core 30 (QLQ-C30)

INTERVENTIONS:
Other: Quality of Life Questionnaire-Core 30 (QLQ-C30) — The HR-QoL evaluation is based on three self-assessment questionnaires distributed to the patients according to the pre-specified data collection schedule. Patients will also complete an additional questionnaire on socio-economic and occupational outcomes
  Other Names: Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13); 5-level EuroQoL EQ5D (EQ5D-5L)

SUMMARY:
OBSTINATE is an observational, national, prospective, multicentric study on Quality of life in patients with unresecable stade III non-small cell lung cancers.

Locally advanced non-small cell lung cancers (NSCLCs with a Tumor, Node and Metastasis [TNM] stage III) patients represent approximately a third of newly discovered NSCLCs every year, and a very heterogeneous group of clinical situations. Therapies are multidisciplinary and very heterogeneous across oncology centers. Patients with locally advanced NSCLC have a high symptom burden that is known to affect their quality of life. Health-related quality of life (HR-QoL) is a specific and multidimensional type of patient-reported outcome (PRO) related to the physical, psychological and social impact of the disease and its treatment as perceived by patients. HR-QoL allows, together with data of efficacy and safety, a more complete assessment of risks and benefits of each treatment. Therefore, QoL maintenance is a valuable consideration for treatment decisions, especially in the rapidly evolving therapeutic landscape of unresectable NSCLC.

The study is designed to collect PROs HR-QoL data from every new patient diagnosed with an unresectable stage III NSCLC over a period of 18 months. We also aim to describe clinical characteristics of these patients, the therapeutic strategies conducted, and outcomes in a "real-word" oncological practice.

DETAILED DESCRIPTION:
OBSTINATE is an observational, prospective, national, multicentric study conducted in patients newly diagnosed with an unresectable stage III NSCLC (with exclusion of early stages NSCLC classified to pathological stage III).

OBSTINATE is a study planned to include 450 patients between 50 to 70 GFPC-affiliates or GFPC-associated centers approximately. All centers are located in France. The participating Site Investigators will be treating physicians within one of the participating centers.

After screening for eligibility checks, patients will receive the Patient Information Note from the Site Investigators. This Patient information Note will describe the study purpose and modalities. Patients who meet the eligibility criteria and do not oppose to data collection will be enrolled. The schedule of the medical visits in the study center will depend on the patient and his/her routine clinical care Protocol-relevant data will be collected by the treating physician within each center, for up to 5 years following the last patient's enrollment in the study.

Patients included in the study will complete the self-assess questionnaires at enrollment and during routine care follow-up, according to pre-specified data collection schedule.

Usual practices or modalities of follow-up of patients will remain unchanged compared to the current clinical practice as the study is designed to provide descriptive summary information.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of NSCLC obtained from a tumor cytology or biopsy
* Treatment-naïve unresectable TNM stage III NSCLC (according to the 8th TNM IASLC edition). Of note, unresectability could be due to either functional limitation or anatomical extension of the tumor.
* Patient willing and able to complete collection of data via self-assessment questionnaires
* Patient without any local or systemic anti-neoplastic treatment are eligible (palliative symptomatic radiotherapy is considered best supportive care)
* Patients participating in other interventional or non-interventional studies can be included.

Exclusion Criteria:

* Early stage NSCLC initially treated locally (surgery or other) and classified as pathological TNM stage III (according to the 8th TNM IASLC edition)
* At the treating physician's discretion, patient not eligible physically or psychologically to be included in a clinical trial
* Inability to read and/or fill out self-assessment questionnaires
* Patient unable to express opposition to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every new patients diagnosed with treatment-naïve unresectable stage III non-small cell lung cancer (according to the 8th TNM IASLC edition).
  Unresectability could be due to either functional limitation or anatomical extension of the tumor.
Sampling Method: Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
QLQ-C30 (defined as the outcomes of a clinical intervention obtained by the patient) | Up to 6,5 years (18 months of recruitment + 5 years). For Cohort 1 & 2, a follow-up post progression is planned
  Change in patient's QLQ-C30 during treatment and follow-up until confirmed progression, loss of follow-up or end of the study compared to Baseline in patients diagnosed with unresectable stage III NSCLC in a "real-world" oncological practice.
  This evaluation is based on self-assess questionnaire distributed to the patients according to pre-specified data collection schedule.
  The primary objective will be addressed in the cohort as a whole, and independently for every cohort of interest.
QLQ-LC13 (defined as the outcomes of a clinical intervention obtained by the patient) | Up to 6,5 years (18 months of recruitment + 5 years). For Cohort 1 & 2, a follow-up post progression is planned
  Change in patient's QLQ-LC13 during treatment and follow-up until confirmed progression, loss of follow-up or end of the study compared to Baseline in patients diagnosed with unresectable stage III NSCLC in a "real-world" oncological practice.
  This evaluation is based on self-assess questionnaire distributed to the patients according to pre-specified data collection schedule.
  The primary objective will be addressed in the cohort as a whole, and independently for every cohort of interest.
EQ5D-5L (defined as the outcomes of a clinical intervention obtained by the patient) | Up to 6,5 years (18 months of recruitment + 5 years). For Cohort 1 & 2, a follow-up post progression is planned
  Change in patient's EQ5D-5L during treatment and follow-up until confirmed progression, loss of follow-up or end of the study compared to Baseline in patients diagnosed with unresectable stage III NSCLC in a "real-world" oncological practice.
  This evaluation is based on self-assess questionnaire distributed to the patients according to pre-specified data collection schedule.
  The primary objective will be addressed in the cohort as a whole, and independently for every cohort of interest.

SECONDARY OUTCOMES:
Baseline demographics | At Baseline
  Stage III unresectable NSCLC patients characteristics: baseline patient demographics at stage III NSCLC diagnosis, clinical, pathological and molecular characteristics (e.g. age, race, comorbidities)
Tumor characteristics as defined by TNM stage | At Baseline
  Characterize the stage III unresectable NSCLC patients by TNM stage according to the 8th TNM IASLC edition
Tumor characteristics as defined by PD-L1 expression status | At Baseline
  Characterize the stage III unresectable NSCLC patients by PD-L1 expression status (tumor propensity score)
Tumor characteristics as defined by mutational status of driver genes | At Baseline
  Characterize the stage III unresectable NSCLC patients by mutational status of driver genes (e.g. epidermal growth factor receptor [EGFR]) anaplastic lymphoma kinase [ALK], reactive oxygen species 1 [ROS1], human epidermal growth factor receptor 2 [HER2], PI3KCA, BRAF, MET, rearranged during transfection [RET], neurotrophic receptor tyrosine kinase [NRTK])
Time from diagnosis to treatment | From date of diagnosis until the date of first documented treatment or start date of best supportive care through study completion, up to 5 year
Modality of follow-up | From date of diagnosis until the date of first documented progression or or date of death from any cause, whichever came first, assessed up to 5 years maximum
  Description of modality of follow-up (e.g. type of imagery used, frequency of medical visit)
Median PFS | From date of first treatment administration up to first documented disease progression and/or death from any cause, whichever came first, assessed up to 60 months
  Time from date of first treatment administration until the date of first documented progression or date to death from any cause, whichever came first as evaluated by investigators.
Median time to progression | From date of first treatment administration up to first documented disease progression and/or death from any cause, whichever came first, assessed up to 60 months
  Time from date of first treatment administration until the date of first documented progression or date to death from any cause, whichever came first as evaluated by investigators.
Median OS (e.g. median PFS, median OS) | From date of first treatment administration up to first documented disease progression and/or death from any cause, whichever came first, assessed up to 60 months
  Time from date of first treatment administration until the date of first documented progression or date to death from any cause, whichever came first as evaluated by investigators.
Treatment characteristics | From date of first treatment administration up to end of study, assessed up to 5 years maximum
  Describe the chemotherapy, radiation therapy and immunotherapy protocols used (e.g. dose, reduction, interruptions, duration)
Best response of treatment | From date of first treatment administration up to end of study, assessed up to 5 years maximum
Duration of response of treatment | From date of first treatment administration up to end of study, assessed up to 5 years maximum
Toxicity of treatment | From date of first treatment administration up to end of study, assessed up to 5 years maximum
  limited to Cohorts 1, 2, 3 and 4 (restricted to significant AEs, which include but are not limited to: serious AEs [SAEs], AEs that led to treatment discontinuation, or any AEs ≥ grade 3 judged clinically significant by the Site Investigator)
Effective treatment compared to initial Multidisciplinary Tumor Board (MDTB) decision | From date of first treatment administration up to end of study, assessed up to 5 years maximum
  Concordance between effective treatment compared to initial MDTB decision
Type of progression (local, loco-regional, metastatic) | At date of first documented progression, assessed up to 5 years maximum
Description of second line of treatment after disease progression | From date of first documented progression up to end of study, assessed up to 5 years maximum
  Treatment characteristics after disease progression including type of treatment (chemotherapy, radiotherapy, immunotherapy or Tyrosine-Kinase inhibitors), treatment duration, stop date of treatment and reason for end of treatment
Change in patients' socio-economic and occupational outcomes using unique self questionnaire | From Baseline, during treatment and follow-up until confirmed progression (of note, for Cohorts 1 and 2, a follow-up post-progression is planned), loss of follow-up or end of the study, assessed up to 5 years maximum
  Change in patients' socio-economic and occupational outcomes during treatment and follow-up until confirmed progression (of note, for Cohorts 1 and 2, a follow-up post-progression is planned), loss of follow-up or end of the study using a dedicated self questionnaire on socio-economic and occupational outcomes
Evaluate the cost-utility of the therapeutic strategy using Quality-Adjusted Life Years (QALYs) | From Baseline, during treatment and follow-up until confirmed progression (of note, for Cohorts 1 and 2, a follow-up post-progression is planned), loss of follow-up or end of the study, assessed up to 5 years maximum

CONTACTS AND LOCATIONS:
Overall Officials: Charles RICORDEL, Principal Investigator — GFPC (Groupe Français de Pneumo-Cancérologie); Christos CHOUAID, Study Director — GFPC (Groupe Français de Pneumo-Cancérologie)
Locations (34):
- France (34):
  - Centre Hospitalier d'Aix en Provence, Aix-en-Provence
  - CHU Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier du Morvan, Brest
  - CHMS, Chambéry
  - Hôpital Paul d'Egine, Champigny-sur-Marne
  - Centre Hospitalier de Chauny, Chauny
  - Centre Hospitalier du Cotentin, Cherbourg
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier d'Elbeuf - Pneumologie, Elbeuf
  - CHD Les Oudairies, La Roche-sur-Yon
  - Hôpital Robert Boulin, Libourne
  - Centre Hospitalier Universitaire DUPUYTREN, Limoges
  - Hôpital du Scorff, Lorient
  - Centre Leon Bérard, Lyon
  - Hôpital Européen, Marseille
  - Hôpital Nord, Marseille
  - Hôpital de Meaux, Meaux
  - Centre Catalan d'Oncologie, Perpignan
  - Centre Hospitalier Intercommunal de Quimper, Quimper
  - CHU Ponchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - CHU La Réunion Site Nord, Saint-Denis
  - Hôpital Privé de la Loire, Saint-Etienne
  - CHU Hôpital Nord, Saint-Etienne
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHU La Réunion Site Sud, Saint-Pierre
  - Institut Lucien Neuwirth, Saint-Priest-en-Jarez
  - CH de Bigorre Tarbes, Tarbes
  - Hôpital d'Instruction des Armées Ste Anne, Toulon
  - CH Bretagne Atlantique, Vannes
  - Centre Hospitalier de Villefranche sur Saone, Villefranche-sur-Saône
  - Centre hospitalier Intercommunal, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No
All collected data that underlie results in a publication